CLINICAL TRIAL: NCT07217730
Title: § PHX-AFK-US: Public Health Exchange Protocol for Anti-Fraud, Kickback Prevention & Secure Chain Integrity in U.S. Healthcare Facilities
Brief Title: Healthcare Integrity & Anti-Fraud Enforcement
Acronym: PHX-AFK-US
Status: Enrolling by invitation | Type: Observational
Sponsor: Truway Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRS-HI-AFK-SC-US-101325-GS
Record Dates: First submitted 2025-10-13; First posted 2025-10-16 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthcare Fraud Schemes; Kickback Networks; Supply Chain Vulnerabilities; Governance Failures; Whistleblower Activation; Regulatory Escalation Pathways; Validator Oversight & DAO Governance; Public Transparency & Auditability
Keywords: Healthcare Integrity; Anti-Fraud; Kickback Prevention; Secure Supply Chain; Validator Governance; Coalition Oversight; NFT Fiscal Instruments; Smart Contract Enforcement; DAO Voting; SHA-256 Notarization; Whistleblower Affidavits; Regulatory Escalation; Public Transparency; Audit Trail; Asset Freeze Logic; CMS / DOJ / OIG Complaints; Procurement Reform; Phantom Billing; Referral Schemes; Medical Device Provenance; Coalition Dashboard; Public Health Exchange; SOP Violations; Facility Sanctions; DeFi Escrow Logic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Flagged Healthcare Facilities - Validator Oversight Cohort: This cohort consists of U.S. healthcare facilities identified through validator affidavits, whistleblower declarations, and coalition intelligence as exhibiting patterns of fraud, kickback schemes, or supply chain vulnerabilities. Facilities are enrolled into the PHX-AFK-US Protocol for prospective observation, reform enforcement, and regulatory escalation. Each facility is subject to smart contract triggers, DAO voting logic, and public dashboard transparency. No biospecimens are retained; all data is notarized via SHA-256 hash anchors and integrated into NFT fiscal declarations and validator ballot modules.
  Interventions: Other: Validator-Governed Reform & Regulatory Escalation Protocol; Device: Coalition-Grade Validator Dashboard Module (CVDM-1); Drug: Coalition-Flagged Pharmaceutical Audit Trigger (CFPAT-1)

INTERVENTIONS:
Other: Validator-Governed Reform & Regulatory Escalation Protocol — This intervention deploys a validator-governed framework to monitor, escalate, and reform healthcare facilities exhibiting fraud, kickback schemes, and supply chain vulnerabilities. It integrates notarized affidavits, smart contract enforcement, NFT fiscal declarations, and DAO voting logic to trigger sanctions, regulatory complaints, and operational restructuring. Facilities are observed prospectively, with all actions logged to a public dashboard and anchored via SHA-256 hash notarization. No biospecimens are retained; all data is legal, technical, and governance-based.
  Other Names: PHX-AFK-US Protocol
Device: Coalition-Grade Validator Dashboard Module (CVDM-1) — The Coalition-Grade Validator Dashboard Module (CVDM-1) is a secure, web-based device deployed across enrolled healthcare facilities to enable real-time validator oversight, whistleblower affidavit intake, and smart contract enforcement. It integrates QR-linked audit trails, NFT fiscal declarations, and DAO voting logic. The device anchors all inputs via SHA-256 hash notarization and transmits reform metrics to coalition dashboards. CVDM-1 supports public transparency, regulatory escalation, and validator governance across the PHX-AFK-US Protocol. It does not collect biospecimens and operates solely within legal, technical, and governance domains.
  Other Names: PHX-AFK-US Governance Terminal
Drug: Coalition-Flagged Pharmaceutical Audit Trigger (CFPAT-1) — The Coalition-Flagged Pharmaceutical Audit Trigger (CFPAT-1) is a governance-based drug intervention targeting facilities with suspected fraud, kickback schemes, or supply chain irregularities involving pharmaceuticals. While not a therapeutic agent, CFPAT-1 functions as a regulatory scaffold that flags drug procurement, formulary manipulation, and referral-linked prescribing patterns. It integrates validator ballots, smart contract logic, and SHA-256 hash anchors to escalate complaints to CMS, DOJ, and state boards. All flagged drugs are traced via QR-linked audit trails and NFT fiscal declarations. No biospecimens are retained; the intervention operates within legal, technical, and governance domains.
  Other Names: CFPAT-1

SUMMARY:
The PHX-AFK-US Protocol is a coalition-backed regulatory scaffold designed to restore healthcare integrity across U.S. facilities. It targets fraud, kickback schemes, and supply chain opacity through validator governance, smart contract enforcement, and public transparency. Anchored by notarized affidavits, NFT fiscal instruments, and dashboard oversight, this protocol empowers whistleblowers, mobilizes validators, and escalates complaints to federal and state regulators. It integrates secure audit trails, DAO voting logic, and asset freeze triggers to ensure accountability, reform, and systemic trust.

DETAILED DESCRIPTION:
The PHX-AFK-US Protocol is a coalition-backed regulatory scaffold designed to restore healthcare integrity across U.S. facilities. It targets fraud, kickback schemes, and supply chain opacity through validator governance, smart contract enforcement, and public transparency. Anchored by notarized affidavits, NFT fiscal instruments, and dashboard oversight, this protocol empowers whistleblowers, mobilizes validators, and escalates complaints to federal and state regulators. It integrates secure audit trails, DAO voting logic, and asset freeze triggers to ensure accountability, reform, and systemic trust.

ELIGIBILITY:
Inclusion Criteria:

Facility has documented billing, compliance, or procurement irregularities.

Facility participates in coalition validator onboarding and SHA-256 protocol enrollment.

Facility provides access to billing, procurement, and whistleblower-anchored datasets for auditing.

Exclusion Criteria:

Facility refuses validator onboarding or coalition integration.

Facility lacks traceable procurement or compliance records.

Facility has no whistleblower declaration or validation artifact.

Facility operates outside U.S. jurisdiction or coalition-recognized governance zones.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of U.S. healthcare facilities identified through coalition-backed validator affidavits and whistleblower declarations. These facilities exhibit patterns of fraud, kickback schemes, and supply chain vulnerabilities. The population is monitored prospectively via smart contract triggers, DAO voting, and public dashboard metrics.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2034-10-13 (Estimated); Study Completion 2034-10-13 (Estimated)

PRIMARY OUTCOMES:
Change in Fraudulent Billing and Kickback Incidents Across Enrolled Facilities | Baseline to 12 Months Post-Validator Onboarding
  Description:
  This outcome measures the change in frequency and severity of fraudulent billing practices-including upcoding, phantom billing, and referral-based kickback schemes-across facilities enrolled in the SHA-256 Trial Protocols.
  Facilities are assessed using the Unified Impact Index derived from:
  Historical billing anomalies
  Validator audit results
  Whistleblower declarations
  SHA-256 hash-anchored incident reports
  Facilities are ranked and monitored for reform compliance, ethical standards, and onboarding validation. All scoring logic is notarized and displayed via coalition dashboards.
  Time Frame: Baseline to 12 Months Post-Validator Onboarding.

SECONDARY OUTCOMES:
Change in Supply-Chain Traceability and Compliance Across Enrolled Facilities | Baseline to 12 Months Post-Validator Onboarding
  This outcome measures change in traceability and regulatory compliance for pharmaceuticals, medical devices, and non-pharmaceutical supplies. Facilities are evaluated using:
  Validator Traceability Score (VTS) composite metrics
  NFT tagging for supply-chain nodes
  Blockchain-based audit trails
  Comparative analysis dashboards identifying gaps and escalation pathways for non-compliant entities

CONTACTS AND LOCATIONS:
Overall Officials: Gavin C Solomon, President & CEO, Principal Investigator — Truway Health, Inc.
Locations (1):
- Truway Health, Inc. , View 34, 401 E 34th Street, S11P, New York, NY 10016, New York, New York, United States